CLINICAL TRIAL: NCT03311113
Title: Pilot Study on the ADherence to Oral Antibiotics in Patients With BONE and Joint Infections (ADABONE)
Brief Title: Adherence to Oral Antibiotics In Patients With Osteoarticular Infections
Acronym: OBSAIO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0467
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Bone and Joint Infection; Adherence, Medication
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with osteoarticular infection: To evaluate drug adherence to oral antibiotic therapy in patients treated for bone and joint infection for a minimum expected duration of 6 weeks.
  Interventions: Other: Drug adherence questionnaire

INTERVENTIONS:
Other: Drug adherence questionnaire — Adherence to oral antibiotic therapy will be assessed by means of a questionnaire adapted from the French standardized self-assessment questionnaire of Girerd et al. This questionnaire has six questions, each question being associated with a score. Patient's drug adherence is classified into three groups based on the total score: of high, moderate and poor adherence. The questionnaire will be carried by a phone call to the patient.

SUMMARY:
Bone and joint infection (BJI) are bacterial infections that can occur after surgery (nosocomial infections) or de novo. They constitute a public health problem in Western Countries . These infections are often difficult to treat, with a high rate of re-hospitalizations (19.5%) caused by relapses or recurrences. The treatment of Bone and joint infection can be surgical and / or pharmacological . Drug treatment is based on the use of parenteral and / or oral antibiotics. It is a curative therapy in most cases, with a prolonged duration ranging from 6 weeks to several months depending on the lesions .

Medication adherence, is a patients' behavior defined as drug intake with optimal attendance and regularity, as prescribed and explained by the physician. It is a key factor in the success of any drug therapy, as drugs don't work in patients who don't take them..

To the knowledge of investigators, there are no published data on the adherence to antibiotic therapy in patients treated for Bone and joint infection. In addition to its prolonged duration, the antibiotic treatment of the Osteoarticular Infections may require several daily drug intakes and may be responsible for severe adverse effects, these three factors being known to adversely affect adherence.

Prevalence, adherence patterns over time and determinants of adherence in this patient population are not known. Currently, drug adherence is not routinely evaluated and is not considered in the treatment of Bone and joint infection in the Regional Center for Complex Bone and joint infection of the investigators.

A specific study evaluating adherence to antibiotic therapy in patients treated for Bone and joint infection appears to be justified.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Affiliation having a social security
* Diagnosis of Bone and joint infections
* Surgical and clinical management of the infection at Hospices Civils de Lyon
* Oral antibiotic therapy prescribed for a minimal duration of six weeks and a defined duration
* Patient's information given and informed consent obtained

Exclusion Criteria:

* Oral antibiotic therapy for Bone and joint infections with no defined duration (chronic therapy)
* Antibiotic therapy for Bone and joint infections administered by parenteral route only
* Patient without a phone number or refusing to communicate by phone
* Patient with physical or mental disability impeding information and consent
* Patient with physical or mental disability impeding communication by phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are prescribed oral antibiotic as a therapy for bone and joint infection for a minimum duration of 6 weeks
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with high, moderate and poor adherence | 3 months
  Adherence will be assessed using a questionnaire adapted from the questionnaire of Girerd et al. with 6 questions. Adherence will be assessed during the antibiotic treatment, after 6 weeks of therapy in all patients included. For the included patients still treated at 3 months, it will be evaluated a second time at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des infections ostéo-articulaires de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No